CLINICAL TRIAL: NCT01656499
Title: Effect of AXOS on the Colon Metabolism in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor Kristin Verbeke, Ph. D., KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ML7245
Record Dates: First submitted 2012-07-30; First posted 2012-08-03 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Gut Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arabinoxylanoligosaccharides (AXOS) (Active Comparator): AXOS (2 x 5g WBE/day)
  Interventions: Dietary Supplement: Arabinoxylanoligosaccharides
- Maltodextrine (placebo) (Placebo Comparator): Maltodextrine (2 x 5g/day)
  Interventions: Dietary Supplement: Maltodextrine

INTERVENTIONS:
Dietary Supplement: Arabinoxylanoligosaccharides
  Arms: Arabinoxylanoligosaccharides (AXOS)
Dietary Supplement: Maltodextrine
  Arms: Maltodextrine (placebo)

SUMMARY:
The purpose of this study is to evaluate the effect of AXOS on parameters of colon metabolism and gut health

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* regular dietary pattern (3 meals/day)
* age: 18-45y
* BMI: 18,5-27 kg/m2

Exclusion Criteria:

* intake of antibiotics 1 month prior to the study
* abdominal surgery in the past, with the exception of appendectomy
* intake of medication influencing the gastro-intestinal system 14 days prior to the study
* in treatment at a dietician
* serious liver- or kidney failure
* vegetarians
* intake of pre- and/or probiotics
* Exposure to radioactivity 1 year prior to the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fecal water toxicity | Participants are followed for 10 weeks, with measurements on 4 specific time points

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven/KU Leuven, Leuven, Vlaams-Brabant, Belgium